CLINICAL TRIAL: NCT03007563
Title: Evaluation of a Smartphone Based Optical Diagnostic Tool for Neonatal Jaundice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); University Hospital, Akershus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014/619
Record Dates: First submitted 2016-12-20; First posted 2017-01-02 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Jaundice, Neonatal; Hyperbilirubinemia, Neonatal
Keywords: Diagnosis; Cell Phones; Infant, Newborn
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia, Neonatal; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- newborn infants checked for jaundice (Experimental): an experimental way of bilirubin concentration estimation from smartphone pictures is applied and compared with two standard methods: bilirubin concentration measured in standard blood samples, and bilirubin concentration measured by transcutaneous device.
  Interventions: Device: bilirubin concentration estimation from smartphone pictures; Procedure: bilirubin concentration measured in standard blood samples; Device: bilirubin concentration measured by transcutaneous device

INTERVENTIONS:
Device: bilirubin concentration estimation from smartphone pictures — pictures taken of the skin covering the breast bone
Procedure: bilirubin concentration measured in standard blood samples
Device: bilirubin concentration measured by transcutaneous device

SUMMARY:
Neonatal jaundice is a common and most often harmless condition. However, when unrecognized it can be fatal or cause serious brain injury. Three quarters of these deaths are estimated to occur in the poorest regions of the world. The treatment of jaundice, phototherapy, is in most cases easy, low-cost and harmless. The crucial point in reducing the burden of disease is therefore to identify then children at risk. This results in the need for low-cost, reliable and easy-to-use diagnostic tools that can identify newborns with jaundice.

Based on previous research on the bio-optics of jaundiced newborn skin, a prototype of a smartphone application has been developed. This prototype will be evaluated in a clinical trial in two hospitals in Norway. A smartphone will be used to take picture of the skin of the newborn, and by using an algorithm an estimate of the bilirubin concentration is made. The results from these estimates will be compared to the bilirubin levels measured in standard blood samples, as well as the results from ordinary transcutaneous measurement devices.

ELIGIBILITY:
Inclusion Criteria:

* born in St.Olavs hospital, Trondheim or in Akershus hospital, Oslo, Norway
* born at term
* normal birth weight

Exclusion Criteria:

* in need of advanced medical treatment

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 342 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Correlation between bilirubin estimates by smartphone pictures and by blood samples | 5 minutes
  Estimate of bilirubin levels from smartphone pictures, compared with bilirubin measurement in blood samples in a correlation study. Correlation will be expressed by Pearson correlation coefficient, r.
Correlation between bilirubin estimates by smartphone pictures and by transcutaneous measurements | 5 minutes
  Estimate of bilirubin levels from smartphone pictures, compared with bilirubin measurements from transcutaneous devices in a correlation study. Correlation will be expressed by Pearson correlation coefficient, r.

CONTACTS AND LOCATIONS:
Overall Officials: Siri Forsmo, md prof, Study Director — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - Akershus University Hospital, Oslo
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aune A, Vartdal G, Bergseng H, Randeberg LL, Darj E. Bilirubin estimates from smartphone images of newborn infants' skin correlated highly to serum bilirubin levels. Acta Paediatr. 2020 Dec;109(12):2532-2538. doi: 10.1111/apa.15287. Epub 2020 Apr 19. PMID 32267569